CLINICAL TRIAL: NCT00564174
Title: A Randomized Controlled Trial Comparing Low Molecular Weight Heparin and Aspirin to Aspirin Alone in Women With Unexplained Recurrent Pregnancy Loss
Brief Title: Low Molecular Weight Heparin and Aspirin in the Treatment of Recurrent Pregnancy Loss: A RCT
Acronym: HepASA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis found no difference in LB rate and lower than expected event rate
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33762; CIHR 37749
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Recurrent Pregnancy Loss; Antiphospholipid Antibody Syndrome
Keywords: recurrent pregnancy loss; lupus anticoagulant; anti cardiolipin antibodies; thrombophilia; low molecular weight heparin; aspirin; randomized clinical trial
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombophilia | interventions — Heparin, Low-Molecular-Weight; Aspirin; Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a (Experimental)
  Interventions: Drug: Low molecular weight heparin and low dose aspirin
- b (Active Comparator): Low dose aspirin only
  Interventions: Drug: Low dose aspirin

INTERVENTIONS:
Drug: Low molecular weight heparin and low dose aspirin — Fragmin 5000 IU/day by subcutaneous injection started at time of randomization and continued until 35 weeks gestation or delivery and low dose aspirin 81 mg/day started pre-conception and continued until 35 weeks gestation or delivery
  Other Names: Fragmin (Dalteparin Sodium); ASA
  Arms: a
Drug: Low dose aspirin — 81 mg enteric coated started pre-pregnancy and discontinued at 35 weeks or delivery
  Other Names: ASA
  Arms: b

SUMMARY:
To compare the livebirth rate of women with recurrent pregnancy loss and autoantibodies randomized to either low molecular weight heparin plus aspirin versus aspirin alone.

DETAILED DESCRIPTION:
Previous studies of these therapeutic regimens in the population of recurrent pregnancy loss and autoantibodies, have not provided conclusive evidence of their efficacy due to small sample size and/or weak study design. We undertook a RCT of low molecular weight heparin plus aspirin versus aspirin alone to investigate if the low molecular weight heparin treatment resulted in an increased rate of livebirths as compared to treatment with aspirin alone.

ELIGIBILITY:
Inclusion Criteria:

* history of two or more unexplained consecutive pregnancy losses prior to 32 weeks
* presence of one of the panel of autoantibodies/thrombophilia markers
* confirmed pregnancy

Exclusion Criteria:

* SLE
* known peptic ulcer disease
* sensitivity to ASA or heparin
* previous thrombotic event
* geographic distance from clinic
* failure to consent

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2000-03; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To investigate whether treatment with LMW heparin plus ASA results in an increased rate of livebirths compared to treatment with ASA alone. | Duration of pregnancy

SECONDARY OUTCOMES:
Secondary outcomes included adverse events and incidence of bone loss in the two groups. | pre-pregnancy through postpartum period

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Laskin, MD, Principal Investigator — Associate Professor, Department of Medicine, University of Toronto
Locations (2):
- Canada (2):
  - McMaster Medical Centre, Hamilton, Ontario
  - Mount Sinai Hosptial, Toronto, Ontario

REFERENCES:
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837